CLINICAL TRIAL: NCT00830765
Title: The Use of Progesterone to Reduce Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, John Morrison, Professor, Ob-Gyn, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-0239
Record Dates: First submitted 2008-12-16; First posted 2009-01-28 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Placebo (Placebo Comparator): The participant will receive a weekly injection of placebo from the time of enrollment up until 34 weeks' gestation or delivery, whichever occurs first.
  Interventions: Drug: Placebo
- Progesterone (Active Comparator): The participant will receive weekly injections of 100mg of OHP17 from the time of enrollment until 34 weeks' gestation or delivery, whichever occurs first.
  Interventions: Drug: Progesterone (OHP17)

INTERVENTIONS:
Drug: Progesterone (OHP17) — 100mg of OHP17 or comparable amount of placebo administered by IM injection weekly until either 34 weeks' gestation or delivery has been achieved, whichever occurs first.
  Arms: Progesterone
Drug: Placebo — 2cc of placebo liquid formulated by pharmacy personnel at the University of Mississippi Medical Center injected IM weekly until 34 weeks' gestation has been reached or delivery, whichever occurs first.
  Arms: 1 Placebo

SUMMARY:
Preterm birth is the most common and costly complication in obstetrics. It complicates up to 11 % of all pregnancies and it is responsible for 70% of sick babies. Recently two studies have shown that giving progesterone (a normal hormone made by the ovaries) prolongs gestation in women who have had a preterm birth in an earlier pregnancy (and therefore are at risk for another early delivery). There are other studies that show that this technique of giving a weekly shot of progesterone does not prevent preterm birth. In addition, There are other groups of patients who are at very high risk for preterm birth which have not been studied. They include: 1.) Cervical cerclage (a stitch in the mouth of the womb); 2.) Multifetal gestation (twins, triplets, etc.); 3.) Women with preterm (<34 weeks) rupture of the membranes; 4.) Women with preterm labor during the current pregnancy with intact membranes who have been tocolyzed (have their labor stopped and are getting ready to go home). We purpose to give weekly shots of progesterone or a placebo in a randomized fashion to women in the first group who are at risk for preterm delivery due to an early birth in a previous pregnancy as well as the other four groups listed. If progesterone given weekly is successful at preventing early delivery as compared to the placebo group then great benefit for these women as well as future pregnancies would be accrued.

DETAILED DESCRIPTION:
A. Introduction Preterm birth occurs in 7-12% of all deliveries, but accounts for over 85% of all perinatal morbidity and mortality.1 Despite many strategies for reducing the incidence of preterm birth none have been totally effective. One treatment that showed promise in earlier small trials was the prophylactic administration of progestational compounds.2,3 However, the reports of efficacy were mixed with some showing benefits4,5 while others did not.6,7 More recently, two randomized clinical trials have shown great promise8,9, and revealed a significant decrease in preterm births among women who received 17 alpha-hydroxyprogesterone caproate (17P)8, or 100mg of progesterone delivered by vaginal suppository per week.9 Indeed support by the American College of Obstetricians and Gynecologists, and March of Dimes as well as others have made this treatment the standard of care in many areas of the country.

The limitations of these studies are that they have small numbers as well as a higher than expected preterm delivery rate among placebo patients. Because of the previous controversy as to the effectiveness of progesterone noted in the 70's - 80's it is incumbent upon other centers to carry out new investigational trials in an effort to confirm their results. Secondly, the studies were limited to singleton pregnancies who were "at risk" for preterm delivery thus not surveying three groups with the highest preterm delivery rate: 1.) Multifetal gestations and cervical insufficiency; 2.) Those who have preterm labor in the current pregnancy that have been tocolyzed; 3.) Women with preterm premature rupture of the membranes.

The purpose of the current study to confirm if possible, the findings of the most recent investigations8,9 using the same patient population and in addition, we will study the effect of progesterone vs placebo in preventing early delivery among multifetal gestations in women who have been diagnosed with preterm labor in the current pregnancy.

B. Specific Aim The aim of this study is to compare progesterone (100mg progesterone weekly) to ascertain if there is a reduction in preterm birth and subsequent neonatal morbidity among patients receiving the active drug. If weekly treatment with this agent can be shown to reduce the incidence of preterm delivery and its surrogate adverse outcomes in the neonate, it will have major impact upon patients and the health care delivery system.

C. Rationale Progesterone as indicated in the Introduction has been shown in some, but not all, studies to reduce incidence of preterm delivery and the adverse effects of prematurity. Progesterone has been shown to reduce the number of oxytocin receptors in the myometrium and be responsible in the near term pregnant women for blocking the onset of labor. Weekly use of this compound, if effective, would be much superior to the tocolytic agents currently available.

D. Benefit to Risk Ratio There is no known harm to mother/fetus/infant of progesterone therapy. This compound has been used in early pregnancies at risk for abortion as well as later in pregnancy to reduce the incidence of prematurity as noted in the Introduction. On the beneficial side, if this treatment proves effective it could prolong pregnancy thus reduce significant neonatal morbidity as well as the emotional cost and expense of such pregnancies.

E. Patient Population Patients will be recruited from the University of Mississippi Medical Center Perinatal Clinics, Antepartum Service and Labor and Delivery area. All patients who meet admission criteria will be offered participation in the study.

F. Materials and Methods Patients seen in the University of Mississippi Perinatal Clinics, Antepartum ward or Labor and Delivery area with preterm labor or who are at risk for preterm labor and who meet other admission criteria (without having exclusion criteria) will be offered participation of this study.

Study Protocol Patients meeting the inclusion criteria will have the study explained to them, including benefits risks and alternative therapy. Patients not desiring to participate in the study will receive our current regimen of preterm birth prevention (observation, risk factor assessment, steroids, progesterone, etc). If they accept inclusion into the study after the above explanation they will be randomized by the use of sequentially numbered, sealed opaque envelopes to either receive progesterone or a placebo injection on a weekly basis. Patients with risk factors for preterm birth (prior preterm birth) will be separately randomized from the multifetal gestations or cervical cerclage and the patients with preterm labor in the current pregnancy as well as preterm rupture of the membranes will also separately randomized (four groups total). Neither patients nor participants will know to which group (placebo vs. progesterone) they are assigned as the pharmacy will keep the randomization schedule and will dispense the two solutions in identical syringes for blinding purposes.

Treatment will begin at different gestational ages dependent upon the four groups noted above. For example, multifetal gestation due to their incidence of labor at earlier gestational ages, will begin treatment at 20 weeks' gestation. Those in the preterm labor with the current pregnancy group or premature rupture of membranes will begin their therapy after admission to the hospital following stabilization. All patients will stop therapy at 34 completed weeks of gestation.

After inclusion into the study, prenatal care will be exactly the same as is our standard for such patients at risk for early delivery with the exception of the weekly administration of the study medicine or placebo. For example, weekly prenatal visits, cervical examinations, ultrasounds, steroids and/or tocolytic treatment (given when preterm labor is diagnosed) will be the same regardless of the group to which the patient is randomized. All groups will have one tube of blood drawn from the placental cord at the time of delivery. There will be no additional visits or costs due to the study itself.

F. Data Analysis Data analysis will be by the standard statistical methodology.

VI. Number of Patients Needed:

A sample size estimation indicates that 320 patients (40 in each of four groups-treatment and placebo) will be necessary to have an 80% power of detecting a significance of < 0.05 in the number of preterm births. It is anticipated that a time period of approximately two years will be needed to enroll this number of participants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy 20 - 34 weeks; cervical dilation <4 cm; risk for preterm birth; multifetal gestation; diagnosis of preterm labor during the current pregnancy effectively tocolyzed); preterm rupture of the fetal membranes (24 - 34 weeks); willing and able to sign Informed Consent Form

Exclusion Criteria:

* Failure to meet inclusion criteria as noted above; contraindication to pregnancy continuation; severe medical diseases such as sickle cell disease with crises, diabetes mellitus (F/R/H), severe preeclampsia etc., (physician judgment; severe fetal/obstetric criteria such as intrauterine growth restriction (<5th percentile, placental abruption,placental previa, etc., (physician judgment); non reassuring fetal assessment; allergy to progesterone compounds; refusal to participate

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2004-06; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Morrison, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Winfred L Wiser Hospital for Women and Infants at the University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Briery CM, Klauser CK, Martin RW, Magann EF, Chauhan SP, Morrison JC. The use of 17-hydroxy progesterone in women with arrested preterm labor: a randomized clinical trial. J Matern Fetal Neonatal Med. 2014 Dec;27(18):1892-6. doi: 10.3109/14767058.2014.892922. Epub 2014 Mar 10. PMID 24512252
- [Derived] Briery CM, Veillon EW, Klauser CK, Martin RW, Magann EF, Chauhan SP, Morrison JC. Women with preterm premature rupture of the membranes do not benefit from weekly progesterone. Am J Obstet Gynecol. 2011 Jan;204(1):54.e1-5. doi: 10.1016/j.ajog.2010.08.022. PMID 20869038

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 Progesterone: The participant will receive weekly injections of 100mg of OHP17 from the time of enrollment until 34 weeks' gestation or delivery, whichever occurs first.
Period: Overall Study
Arm/Group | 1 Placebo | 2 Progesterone
Started | 73 | 71
Completed | 70 | 69
Not Completed | 3 | 2
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Placebo | 2 Progesterone | Total
Number analyzed (Participants) | 73 | 71 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 71 | 144
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.0) | 23.3 (5.8) | 24.4 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 71 | 144
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 71 | 144

OUTCOME MEASURES:

1. Primary Outcome: Weeks Gestation at Birth Among Patients Receiving the Active Drug.
Description: Weeks gestation at birth, the interval to delivery, or neonatal morbitity.
Time Frame: Through delivery, until discharge up to 40 weeks gestation
Population: Intention to treat analysis in both groups
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- Progesterone Group; Placebo Group: Progesterone injection was compared to placebo injection on a weekly basis.
Arm/Group | Progesterone Group | Placebo Group
Number analyzed (Participants) | 71 | 73
weeks | 31.9 (3.5) | 30.2 (3.1)

ADVERSE EVENTS:
Arm/Group | 1 Placebo | 2 Progesterone
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/71
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No